CLINICAL TRIAL: NCT02921802
Title: Revlimid 5 mg Capsules Special Use-results Surveillance (All-case Surveillance)
Brief Title: A Study of Special Use Results Surveillance of Revlimid 5mg Capsules
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-Celgene-JP-PMS-001a
Record Dates: First submitted 2016-09-30; First posted 2016-10-03 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma; Myelodysplastic Syndromes
Keywords: Teratogenicity; Thrombocytopenia and haemorrhage; Neutropenia and infection; Venous thromboembolism; Allergic reactions; Diarrhoea or constipation; Peripheral neuropathy; Cardiac failure; Arrhythmia; Renal failure; Myocardial infarction; Interstitial lung disease; Tumour lysis syndrome; Transformation from myelodysplastic syndrome to acute myeloid leukemia
MeSH Terms: conditions — Multiple Myeloma; Myelodysplastic Syndromes; Teratogenesis; Thrombocytopenia; Hemorrhage; Neutropenia; Infections; Venous Thromboembolism; Hypersensitivity; Diarrhea; Constipation; Peripheral Nervous System Diseases; Heart Failure; Arrhythmias, Cardiac; Renal Insufficiency; Myocardial Infarction; Lung Diseases, Interstitial; Tumor Lysis Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who received Revlimid: Among relapsed or refractory multiple myeloma and Myelodysplastic syndrome (MDS) with a deletion 5q cytogenetic abnormality patients, all patients who received Revlimid will be targeted in this surveillance.

SUMMARY:
To understand the safety and efficacy of Revlimid® 5 mg Capsules (hereinafter referred to as Revlimid) in all patients who are treated with it under the actual condition of use pursuant to the conditions of approval.

1. Planned registration period This period started on the date of initial marketing of Revlimid and will end at the time when the planned number of patients to be enrolled is reached.
2. Planned surveillance period This period started on the date of initial marketing of Revlimid and will end on the day when the approval condition related to all-case surveillance is terminated.

ELIGIBILITY:
Inclusion Criteria:

* Among relapsed or refractory multiple myeloma and Myelodysplastic syndrome (MDS) with a deletion 5q cytogenetic abnormality patients, all patients who received Revlimid will be targeted in this surveillance.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among relapsed or refractory multiple myeloma and Myelodysplastic syndrome (MDS) with a deletion 5q cytogenetic abnormality patients, all patients who received Pomalyst will be targeted in this surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 4626 (Actual)
Dates: Start 2010-07-20 (Actual); Primary Completion 2013-03-29 (Actual); Study Completion 2013-03-29 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to 6 months
  Number of participants with adverse events for 6 month treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Shinko Hospital, Kobe, Hyōgo, Japan